CLINICAL TRIAL: NCT07390968
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Controlled Trial of the Safety and Immunogenicity of a Self-Amplifying mRNA COVID-19 Vaccine in Adult Hematopoietic Cell Transplant Recipients
Brief Title: Self-Amplifying mRNA COVID-19 Vaccine (LUNAR-COV19) Versus Comirnaty Vaccine in Adult Hematopoietic Cell Transplant Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Arcturus Therapeutics, Inc. (Industry); Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1125827; NCI-2026-00148 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20962 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded to the treatment assignment, All investigative study center personnel involved in participant evaluations will remain blinded to the treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (LUNAR-COV19) (Experimental): Patients receive LUNAR-COV19 IM on days 1, 29 and 113 in the absence of medical conditions or unacceptable toxicity. Additionally, patients undergo nasal swab at screening and at time of suspected SARS-CoV-2 infection, as well as blood sample collection throughout the study.
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine ARCT-021; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration
- Arm II (Comirnaty) (Experimental): Patients receive SARS-CoV-2 Comirnaty IM on days 1, 29 and 113 in the absence of medical conditions or unacceptable toxicity. Additionally, patients undergo nasal swab at screening and at time of suspected SARS-CoV-2 infection, as well as blood sample collection throughout the study.
  Interventions: Biological: Tozinameran; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA Vaccine ARCT-021 — Given IM
  Other Names: ARCT 021; ARCT-021; ARCT-021 COVID-19 Vaccine; ARCT-021 SARS-CoV-2 Vaccine; ARCT021; LUNAR-COV19
  Arms: Arm I (LUNAR-COV19)
Biological: Tozinameran — Given IM
  Other Names: BNT 162b2; BNT-162b2; BNT1162b2 SARS-CoV-2 Vaccine; BNT162b2; BNT162b2 (Pfizer-BioNTech); BNT162b2 COVID-19 Vaccine; Comirnaty; Pfizer COVID-19 Vaccine; Pfizer-BioNTech COVID-19 Vaccine; Pfizer/BioNTech COVID-19 Vaccine; SARS-CoV-2 SP mRNA LNP Vaccine BNT162b2
  Arms: Arm II (Comirnaty)
Procedure: Biospecimen Collection — Undergo nasal swab and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase IIb trial compares the effect of LUNAR-COV19 vaccine to Comirnaty vaccine in treating adult patients who have received a hematopoietic cell transplant (HCT). Guidelines recommend repeating severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) vaccination of 3 messenger ribonucleic acid (mRNA) vaccines followed by a fourth booster 3-6 months after treatment. However, vaccination is less effective in HCT patients compared to healthy people due to impaired immune responses. LUNAR-COV19, a self-amplifying mRNA vaccine, may help the body's own immune system recognize the SARS-CoV-2 spike protein and fight the virus by using a special mRNA that copies itself for a stronger response. Vaccines made from mRNA with SARS-CoV-2, such as Comirnaty, may help the body build an effective immune response. This may provide active protection against SARS-CoV-2 infection. LUNAR-COV19 may be safe and tolerable and may generate a better and more durable immune response than the Comirnaty vaccine in adult patients who have received a HCT.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive LUNAR-COV19 intramuscularly (IM) on days 1, 29 and 113 in the absence of medical conditions or unacceptable toxicity. Additionally, patients undergo nasal swab at screening and at time of suspected SARS-CoV-2 infection, as well as blood sample collection throughout the study.

ARM II: Patients receive SARS-CoV-2 Comirnaty IM on days 1, 29 and 113 in the absence of medical conditions or unacceptable toxicity. Additionally, patients undergo nasal swab at screening and at time of suspected SARS-CoV-2 infection, as well as blood sample collection throughout the study.

After completion of study treatment, patients are followed up at days 115, 120, 127, 141 and 281.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent (where locally approved)
* Have received an allogeneic HCT within the prior 365 days
* Have no relapse or progression of underlying malignancy
* Have platelets ≥ 30,000/mm^3
* Not pregnant (confirmed with negative urine or serum pregnancy test, if applicable)
* Willingness to take study vaccine and complete necessary study procedures
* If of childbearing potential, must agree to use a highly effective method of birth control or abstain from heterosexual activity for the course of the study through at least 60 days after the last dose of the study vaccine

Exclusion Criteria:

* Current infection with SARS-CoV-2 or infection within the prior 28 day period
* Positive for SARS-CoV-2 by nasal swab polymerase chain reaction (PCR) at screening
* Currently receiving any approved, authorized, or investigational direct-acting antiviral drug against SARS-CoV-2
* Received any approved, authorized, or investigational monoclonal anti-SARS-CoV-2 antibody therapy within the prior 180 days before screening
* Received a SARS-CoV-2 vaccine after HCT or within 28 days prior to HCT
* Participation in any other concurrent clinical trial of an experimental treatment or prevention for SARS-CoV-2
* Receiving > 1 mg/kg/day corticosteroids within the prior 7 days
* Active infection that is not adequately controlled, as determined by the investigator
* Have received therapies that cause profound T-cell or B-cell depletion within 30 days of enrollment, or anticipated to receive such therapies within 3 months of enrollment
* Have received immunoglobulin replacement therapy (IGRT) within 30 days of enrollment, or anticipated to receive IGRT within 3 months of enrollment
* Have a history of suspected or documented myocarditis or pericarditis
* Any inability to take study vaccine or comply with study procedures that, in the opinion of the investigator, would make the participant unsuitable for the study
* Individuals with a known history of severe hypersensitivity reactions, including anaphylaxis, or other significant adverse reactions to any vaccine or any vaccine excipient. Have any other condition that would, in the investigator's judgment, contraindicate participation in the clinical study due to safety concerns with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of neutralizing antibody (nAb) against spike protein matching the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) variant | At 28 days after the third vaccine dose, assessed up through day 141
  Will compare log10-transformed SARS-CoV-2 nAb titers at 28 days following the third vaccination (day 141) between study arms using linear mixed effects models with fixed effects for time points when nAb titers are measured up until day 141 (days 29, 113, and 141; baseline as the reference category), study arm, the interaction between time points and study arm, and stratification variables (time since hematopoietic cell transplantation [HCT] and site). Subject-specific random effects will be included. Model estimates will be exponentiated and presented as a ratio of GMTs, with 90% confidence intervals, to correspond with the two-sided alpha of 0.10 used for power calculations.

SECONDARY OUTCOMES:
Percentage of participants with one or more solicited local or systemic reactogenicity signs and symptoms | For up to 7 days following each vaccination
  Will tabulate the number and severity of solicited local or systemic reactogenicity signs and symptoms overall and by randomization group. Will compare the probability of at least one solicited local reaction or systemic adverse event after each vaccination dose by randomization arm using generalized linear mixed effects models, with logit link, similar to the models described for the seroresponse outcome.
Percentage of participants with unsolicited adverse events (AEs) | Up to 28 days following each vaccination
  Will tabulate the number and severity of unsolicited AEs overall and by randomization group. Will also report the number and percentage of participants with at least one of each of these types of AEs, by dose, severity, and study arm. The probability of at least one unsolicited AE will be compared between study arms using similar models.
Percentage of participants with one or more serious AEs, or AEs of special interest (AESIs) | Following first study vaccine dose until 6 months following last vaccination
  Will tabulate the number and severity of serious AEs or AESIs overall and by randomization group. Will also report the number and percentage of participants with at least one of each of these types of AEs, by dose, severity, and study arm. The probability of at least one serious AE or AESI will be compared by study arms using time-to-event methods.
nAb GMT against spike protein matching the SARS-CoV-2 variant included in the vaccine | At 28-84 days after each vaccine dose, and at 6 months after the last dose
Anti-spike immunoglobulin G GMT against Spike protein matching the SARS-CoV-2 variant included in the vaccine | At 28-84 days after each vaccine dose, and at 6 months after the last dose
Seroresponse rates | At 28-84 days after each vaccine dose, and at 6 months after the last dose
  Will be defined as the proportion of participants with a 4-fold or greater increase in nAb titers. Will be compared by study arm using mixed effects models, but with a binomial distribution and logit link, and using the baseline nAb as a covariate rather than a dependent variable. Comparisons from these models will be presented as odds ratios with 95% confidence intervals. Per-protocol (PP) analyses among the PP cohort may be performed as a sensitivity analysis.
Quantitative levels of anti-Spike T cell responses | At 28-84 days after each vaccine dose, and at 6 months after the last dose
  Will be based on a validated intracellular cytokine staining assay demonstrating interferon-γ, interleukin-2, or both.
New events of late-acute or chronic graft-versus-host disease (GVHD) of grade 3 or higher | Up to day 141
  Will compute the cumulative incidence of late-acute or chronic GVHD of grade 3 or higher by randomization arm using time-to-event methods.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hill, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No